CLINICAL TRIAL: NCT02638233
Title: Direct Observed Therapy With Ledipasvir/Sofosbuvir in Treatment-naïve Patients With Chronic Genotype 1 HCV (Hepatitis C Virus) Infection Receiving Opiate Substitution Therapy
Brief Title: Therapy With Ledipasvir/Sofosbuvir in Patients With Genotype 1 HCV Infection Receiving Opiate Substitution Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wilhelminenspital Vienna (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Michael Gschwantler, Prof.Dr, Wilhelminenspital Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIL4ME2015/01
Record Dates: First submitted 2015-10-05; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Hepatitis C
Keywords: CHC; IVDA (intravenous drug abuse); Hepatitis C; Sofosbuvir; Ledipasvir; Opiate Substitution Therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Substance Abuse, Intravenous; Hepatitis C | interventions — Sofosbuvir; ledipasvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sofosbuvir 400mg/Ledipasvir 90 mg (Other): Subjects will receive sofosbuvir 400mg q.d p.o and ledipasvir 90 mg q.d p.o (FDC) for 8 weeks
  Interventions: Drug: Sofosbuvir 400mg / Ledipasvir 90 mg (FDC)

INTERVENTIONS:
Drug: Sofosbuvir 400mg / Ledipasvir 90 mg (FDC)
  Other Names: Harvoni

SUMMARY:
Patients with chronic hepatitis C that are under opiate substitution therapy are likely to have psychiatric comorbidities such as depression; hence an Interferon based therapy is contraindicated. Additionally many of these patients have a borderline compliance, which makes it impossible to treat them at specialized hepatological centers. An ideal opportunity to treat this patients is treatment with DAAs (Direct Acting Antiviral) which can be administered daily together with the opiate substitution therapy at a low threshold facility.

DETAILED DESCRIPTION:
Background:

Patients with active or previous i.v.-drug abuse and patients receiving opiate substitution therapy (OST) represent a major subgroup of the patients with chronic hepatitis C (CHC). Till some years ago it was held, that patients with a history of i.v.-drug abuse and patients receiving OST should not be considered for interferon-based antiviral treatment because of their poor compliance. However, during the past years it became clear, that patients on OST who are considered to be stable by their physicians are good candidates for antiviral therapy. Several studies have shown that SVR (sustained virological response rates) achieved in these patients are similar to results in patients without a history of i.v. drug abuse.

Subgroups of patients receiving OST:Patients receiving OST represent a very heterogeneous population. However, based on empirical observation of the behavior/compliance of each individual patient they can be assigned to one of the following three groups:

Group 1: Patients with very good compliance. These patients do not take drugs anymore and demonstrate a very good compliance. If anti HCV therapy is indicated, these patients can be referred to and treated at a hepatologic Center (i.e. hospital). Such patients have been included in various phase III trials of new direct acting antiviral agents (DAAs).

Group 2: Patients with a very poor compliance. These patients do not keep appointments (regardless whether it is at a low threshold facility or at a hospital). Due to their lack of compliance antiviral therapy of these patients is not feasible.

Group 3: Patients with a borderline compliance. These patients do come to a low threshold facility on a daily basis where they get OST under direct observation of a physician or a nurse. These patients are reluctant to go to specialized hepatitis centers (high inhibition threshold) and hence cannot be treated there. However, anti-HCV treatment can be applied together with OST under direct observation of a physician or a nurse at the low threshold facilities. The "Ambulatorium Suchthilfe Wien" a "low threshold facility" (LTF): The "Ambulatorium Suchthilfe Wien" is a facility that offers medical care to patients with active or former i.v. drug abuse (= (ex-)PWIDs). The medical team at these low-threshold facilities (=LTFs) includes general practitioners, specialists in internal medicine, psychiatrists and nurses. In contrast to hospitals (hepatologic centers in Austria with outpatient clinics in a large hospital), where there is a relatively high "psychological" inhibition threshold for PWIDs with CHC, the LTFs are located in "normal" houses. The setting is such that the "psychological" inhibition threshold for PWIDs to go there is low. At the LTFs (ex-)PWIDs can obtain OST on a daily basis under direct observation of a physician or a nurse. Hence, the patients have a high motivation to come to these facilities daily (to avoid withdrawal symptoms - they do not have a similar incentive/interest/motivation to go to a hospital on a regular basis). The direct observed OST prevents potential selling of medication on the black market. Anti-HCV treatment at the "Ambulatorium Suchthilfe Wien":

Univ.-Prof. Dr. Michael Gschwantler, an experienced hepatologist is cooperating with the "Ambulatorium Suchthilfe Wien" (=LTF). He visits the facility at least once a week (and immediately in the case of any serious problem) and takes care of the patients with regards to hepatitis/liver diseases. Prof. Gschwantler does this voluntarily and unsalaried. He performs routine laboratory and sonographic evaluation of the liver directly at the LTF. Prof. Gschwantler has already treated a small number of eligible "group 3 patients" (patients with borderline compliance as described before) with interferon-based treatment directly at the LTF (patients didn't need to go to a hospital). However, beside compliance issues contraindications against interferon (e.g. due to depression) prevent many (ex-)PWIDs from being treated at the moment.

Study drug:

In this non-interventional study patients with chronic hepatitis C, genotype 1, will be treated with Harvoni® (Sofosbuvir/Ledipasvir). Harvoni® has been approved for treatment of chronic hepatitis C. For treatment-naïve patients with genotype 1 infection without liver cirrhosis the recommended duration of treatment is 8 weeks. In this non-interventional study treatment with Harvoni® will be performed exactly according to the label.

The study drug will kindly be provided by Gilead.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 1 HCV infection
* Fibrosis F0-F3 (i.e. non-cirrhotic confirmed by Fibroscan <12.5kPa)
* Stable opiate substitution therapy
* Regular visits at the low threshold facility during the last month

Exclusion Criteria:

* Lack or unwillingness of safe contraception, pregnancy
* Liver cirrhosis (Fibroscan ≥12.5kPa)
* Coinfection with HBV (Hepatitis B Virus) or HIV (coinfection with HIV is excluded only because there are very few coinfected patients under care at the "Ambulatorium Suchthilfe Wien" and hence this subpopulation would be very small)
* Severe comorbidities resulting in a life expectancy of less than five years
* HCC (Hepatocellular carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of pills taken during the treatment phase will be calculated as a parameter for adherence to therapy for each individual subject. | 8 Weeks
  Study drugs will administered daily together with the opiate substitution therapy under the supervision of qualified site personnel and recorded on a worksheet for each subject. At the end of the treatment phase, the total number of DAA pills taken will be assessed as percentage for each subject and for the whole study population.

SECONDARY OUTCOMES:
Sustained Virologic Response (SVR) 12 Weeks after End of Therapy (SVR 12) | 12 Weeks after end of Therapy
  Viral load will be measured via PCR 12 Weeks after the End of Therapy
Sustained Virologic Response (SVR) 24 Weeks after End of Therapy (SVR 24) | 24 Weeks after end of Therapy
  Viral load will be measured via PCR (polymerase chain reaction) 24 Weeks after the End of Therapy
Safety and tolerability (total number of observed adverse events) | 20 weeks
  Safety and tolerability of Ledipasvir/Sofosbuvir in patients with chronic hepatitis C under opiate substitution therapy at a low threshold facility will be assessed by reporting total number of adverse event and laboratory abnormalities observed in each patient. Total number of observed adverse events and laboratory abnormalities will be reported tabulated by body system. Adverse events will be observed during the 8 weeks treatment phase and the 12 week follow up phase, for a total duration of 20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gschwantler, Prof. MD, Principal Investigator — Wilhelminenspital Vienna
Locations (1):
- Wilhelminenspital, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Schutz A, Moser S, Schwanke C, Schubert R, Luhn J, Gutic E, Lang T, Schleicher M, Haltmayer H, Gschwantler M. Directly observed therapy of chronic hepatitis C with ledipasvir/sofosbuvir in people who inject drugs at risk of nonadherence to direct-acting antivirals. J Viral Hepat. 2018 Jul;25(7):870-873. doi: 10.1111/jvh.12857. Epub 2018 Feb 6. PMID 29316001